CLINICAL TRIAL: NCT04311892
Title: Hip Abductor Muscle Dysfunction After Nailing of Proximal Femoral Fractures, Incidence and Contributing Factors.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ahmed Adel Khalifa, Assistant professor orthopaedic and traumatology, Principal Investigator, Clinical Professor, South Valley University
Other Study IDs: 1
Record Dates: First submitted 2019-01-14; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: EMG of the hip abductor muscles — EMG will be carried out to examine the (superior gluteal nerve) SGN for all patients. The muscles will be evaluated according to the criteria of the American Academy of Electrophysiological Medicine for needle EMG. In order to exclude patients with polyneuropathy, radiculopathy, or plexopathy, nerve conduction studies of both lower extremities will be performed. Then, gluteus medius muscles will be assessed bilaterally to evaluate the SGN, the vastus medialis muscle for L4 root, tibialis anterior muscle for L5 root, and gastrocnemius muscle for S1 root.

SUMMARY:
Proximal femoral fractures(PFFs) are common with advancing age. Proximal femoral nail (PFN) is now increasingly used to fix unstable fractures. Studies have demonstrated that muscle strength deficit is significantly large after PFFs. N. Ivanova et al found that hip muscle isometric strength for the fractured leg was significantly decreased 1 week and 6 months postoperatively. Besides, a recent study done by Nitin Wale et al concluded that abductor weakness and trendeleburg gait are fairly common in patients treated with PFN and this complaint is often overlooked. Despite significant improvement in muscle function after at least 6 months of physiotherapy as demonstrated by previous studies, we didn't come over a study explaining the main causes of remaining abductor lurch in patients with united fracture of the proximal femur treated using proximal femoral nail (short type).

DETAILED DESCRIPTION:
In a group of patients treated at our hospital for fracture of the proximal femur using different generations of the proximal femoral nail and after full fracture union, although they had an excellent hip function we noticed that the majority of the patients still suffering from limping and abductor lurch with a Trendelenburg gait.

Purpose: to detect hip abductor muscle dysfunction after treating proximal femoral fracture using a proximal femoral nail (short type)

Research Questions: what is the reason(s) for remaining abductor lurch in patients with proximal femoral fracture treated with PFN?

Study Design: an observational retrospective

Study Group number: 20 patients (to be modified according to the number of patients registered at the study setting)

Assessment: (will be measured on both operated and non-operated sides)

* Clinical:

  1. Harris hip score.
  2. Leg length discrepancy: measured as the true length from the ASIS to the medial malleolus.
  3. The bulk of the abductor musculature: measured as the distance between the ASIS anteriorly and the ischial tuberosity posteriorly.
  4. Trendelenburg gait: assessed using modified McKay criteria2. These criteria measure pain symptoms, gait pattern, Trendelenburg sign status, and the range of hip joint movement
* Radiological:

  1. Fracture union: assessed using Apley and Solomon's criteria6. Complete bone union according to these criteria is defined as the time at which there is no pain upon local palpation, no swelling in the limb, ability to walk without support and pain-free, and evidence of a radiographic bridging callus or trabecula between fragments.
  2. Neck shaft angle: as the angle between the neck axis and the anatomical axis of the proximal femur.
  3. Leg length discrepancy: as the distance between a fixed reference point on the lesser trochanter on both sides and the trans-ischial line.
  4. Amount of nail prominent from the greater trochanter.
  5. Hip horizontal offset: the length of a line drawn from the centre of the femoral head and perpendicular to the anatomical axis of the femur.
* Neurophysiological:

EMG will be carried out to examine the (superior gluteal nerve) SGN for all patients. The EMGs will be performed by the same neurophysiologist. The muscles will be evaluated according to the criteria of the American Academy of Electrophysiological Medicine for needle EMG. In order to exclude patients with polyneuropathy, radiculopathy, or plexopathy, nerve conduction studies of both lower extremities will be performed. Then, gluteus medius muscles will be assessed bilaterally to evaluate the SGN, the vastus medialis muscle for L4 root, tibialis anterior muscle for L5 root, and gastrocnemius muscle for S1 root. First, resting activities will be assessed for the signs of acute denervation (fibrillation and positive sharp waves), followed by observation of the recruitment pattern examination of the motor unit action potential (MUAP) amplitudes, and time characteristics. Finally, motor patterns of interferences will be investigated during muscle contractions to obtain information about denervation and reinnervation of examined muscles

Outcomes to be measured:

* Primary outcome: Neurophysiological status of Hip abductors function (EMG)
* Secondary outcome: HHS, altered radiological hip biomechanics

ELIGIBILITY:
Inclusion Criteria:

* patients treated with this type of implant for proximal femoral fracture with or without abductor lurch, follow up more than 6 months, fracture full union

Exclusion Criteria:

* patients suffering from neurological disorder affecting the same side of surgery (polio- hemiplegia), less than 6 months follow up, fracture non- or delayed union, polytraumatized patients, pathological fractures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patients (male or females) treated in our hospital for fracture of the proximal femur with or without obvious abductor lurch
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Hip abductor muscles neuro-physiological state | 4 months
  the state of the hip abductor muscles regarding it innervation and the state of the muscle fibers itself

SECONDARY OUTCOMES:
proximal femoral shortening | 4 months
  shortening of the treated side measured on the AP radiograph

CONTACTS AND LOCATIONS:
Locations (1):
- Qena university hospital, South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided